## Study Title: Improving Future Thinking Among Mothers to Reduce Harsh Parenting and Improve Child Outcomes

NCT #: NCT05229146

Statistical Analysis Plan

10 September 2024

Dr. Julia Felton



Research Administration Henry Ford Health System 1 Ford Place – 2F Detroit, MI 48202-2689 (313) 874-4464 Office (313) 874-4288 Fax

## **EXPEDITED AMENDMENT APPROVAL LETTER**

**To:** Julia Felton, Ph.D.

Center for Health Policy and Health Services Research

**From:** Jonathan K Ehrman, Ph.D.

Date: September 10, 2024

**IRB No.:** 15407

Title: The Parent-Child Memory Study: Improving Future Thinking among Mothers from a

Traditionally Underserved Community to Reduce Harsh Parenting and Improve Child

Outcomes.

Study

December 28, 2023

Approval Date:

Amendment September 04, 2024

Approval Date:

Amendment Other-New Statistical Analysis Plan

**Description:** 

The modification to your study was reviewed and approved by the Henry Ford Health IRB via expedited review on September 04, 2024.

The IRB determined that the Criteria for IRB **approval** are met pursuant to 45 CFR 46.111 and if applicable, 21 CFR 56.111. The following changes/documents have been approved:

Statistical Analysis Plan (Misc/Other)

Any revisions to the protocol must be submitted to the IRB for review and approval prior to implementation. Please contact the IRB Administration Office at IRBQuestions@hfhs.org if you have any questions or concerns.

## **Data Analytic Plan**

Primary Outcomes: Changes in delay discounting and consideration of future consequences.

Descriptive statistics will be used to characterize the sample and psychometric properties will be examined (reliability, etc.). Changes in quantitative measures (including Monetary Choice Questionnaire and Consideration of Future Consequences Scale – adapted for parenting) will be examined in a number of ways. First, we will examine each variable to evaluate mean, standard deviations, skew and kurtosis. We will examine the overall number of mothers who demonstrated decreases in delay discounting (5-Trial Adjusting Measure of Delay Discounting). We will use a *t*-test to examine differences in mean levels of consideration of future consequences (Consideration of Future Consequences Scale-Parenting). We will set statistical significance at *p*<.05.

Secondary Outcomes: Changes in parent-child behaviors, parenting, child emotion regulation, and evaluation of client satisfaction.

Descriptive statistics will also be examined for all secondary outcomes. We will then evaluate changes in our measures of parent-child behavior (using the Dyadic Parent-Child Interaction Coding System), parent-reported parenting (using the Alabama Parenting Questionnaire), and child emotion regulation (using the Emotion Regulation Checklist) using t-tests and RCIs. We will set statistical significance at p<.05. We will also examine overall mean scores on a measure of participant satisfaction (the adapted Client Satisfaction Questionnaire).